CLINICAL TRIAL: NCT05027152
Title: Correlation of "Myositis Functional Index-3 (Fi-3)" With Muscle Function Assessed by Isokinetic Dynamometry and Effects of Repetitive Task Training in Patients With Inflammatory Myopaties
Brief Title: Muscle Function and Effects of Repetitive Task Training in Patients With Inflammatory Myopaties
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Espirito Santo (Other)
Responsible Party: Principal Investigator, Samira Tatiyama Miyamoto, PhD, Professor, Federal University of Espirito Santo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUEspiritoSanto
Record Dates: First submitted 2021-07-29; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Idiopathic Inflammatory Myopathy; Dermatomyositis; Polymyositis
Keywords: exercise; muscle function; functional capacity; quality of life
MeSH Terms: conditions — Myositis; Dermatomyositis; Polymyositis; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Group 1: Traditional resistance exercises. Group 2:The repetitive task training group
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional resistance exercises (Experimental): The resistance training group will perform traditional resistance exercises with an intensity of 30%-60% of a voluntary repetition maximum and 1 to 2 sets of 10 repetitions each exercise.
  Interventions: Other: Resistance training
- repetitive task training (Experimental): The repetitive task training group will carry out exercises involving upper and lower limbs.
  Interventions: Other: Repetitive task training

INTERVENTIONS:
Other: Resistance training — The resistance training group will perform traditional resistance exercises with an intensity of 30%-60% of a voluntary repetition maximum and 1 to 2 sets of 10 repetitions each exercise. The repetitive task training group will carry out exercises involving upper and lower limbs.
  Arms: traditional resistance exercises
Other: Repetitive task training — The repetitive task training group will carry out exercises involving upper and lower limbs.
  Arms: repetitive task training

SUMMARY:
Idiopathic inflammatory myopathies lead to important functional limitations resulting from the loss of muscle strength and endurance, especially in the hip and shoulder, which leads to a significant loss of quality of life for patients. The aim of this study is to correlate the "Myositis Functional Index-3 (FI-3)" with muscle function assessed by computerized isokinetic dynamometry, electromyography and magnetic resonance through an observational study; and to compare the effects of a repetitive task training program with a resistance exercise program through an interventional study in patients with inflammatory myopathies. It is expected that FI-3 will present a good correlation with muscle function assessed by computerized isokinetic dynamometry and electromyography, given its reduced cost and less time spent on evaluation. It is also expected to demonstrate that repetitive task training is as efficient and safe as resistance exercises.

DETAILED DESCRIPTION:
Idiopathic inflammatory myopathies lead to important functional limitations resulting from the loss of muscle strength and endurance, especially in the hip and shoulder, which leads to a significant loss of quality of life for patients. PURPOSE: to correlate the "Myositis Functional Index-3 (FI-3)" with muscle function assessed by computerized isokinetic dynamometry, electromyography and magnetic resonance through an observational study; and to compare the effects of a repetitive task training program with a resistance exercise program through an interventional study in patients with inflammatory myopathies. METHODS: this is an observational cross-sectional study for the observational study and an interventional study/randomized clinical trial for the interventional study. The study will be held at the Cassiano Antônio de Moraes University Hospital (HUCAM) and at the Interprofessional Health Clinic (CEIS) of the Federal University of Espírito Santo (UFES), located in the city of Vitória, Espírito Santo. Patients will come from the Rheumatology Service of HUCAM For the observational study, 30 patients with inflammatory myopathies and 15 healthy individuals matched for age and sex. For the interventional study, the 30 patients evaluated in the observational study will be randomized into two intervention groups. To participate in the research, patients must have a diagnosis of polymyositis or dermatomyositis (Bohan and Peter criteria); age ≥18 years; duration of disease since diagnosis for more than six months; stable medication ≥3 months; chronic inactive or mildly active but stable myositis for at least 3 months prior to observation; HAQ≥0.5. They may not have serious cardiac or pulmonary conditions; severe osteoporosis; unable to exercise; neoplasm; cognitive disorders; and acute or chronic infection. Healthy individuals must be age and sex matched with patients and may not have severe cardiac or pulmonary conditions; severe osteoporosis; unable to exercise; neoplasm; cognitive disorders; and acute or chronic infection. Patients will be evaluated in two moments: before starting the training programs and after 12 weeks. Healthy individuals will be evaluated only once. The data from the evaluations carried out before starting the training programs will be used for the analysis of the observational study. Participants will be evaluated for variables: muscle endurance (Functional Index-3 and isokinetic dynamometry), muscle strength (Manual Muscle Test 8 and isokinetic dynamometry), muscle activation (electromyography), muscle damage (magnetic resonance imaging of thigh muscles), cardiopulmonary capacity (6-minute walk test), pain (visual analogue scale), functional capacity (Health Assessment Questionnaire), quality of life (SF-36), disease activity (PGA, SGA, MDAAT, creatine phosphokinase and aldolase) and disease damage (MDI). In addition, demographic and clinical data such as date of birth, age, sex, self-reported race-color, marital status, occupational status, weight, height, date of first symptoms, date of diagnosis, comorbidities and medications in use will also be collected. The training program will last 12 weeks, twice a week in person with the supervision of physiotherapists and once a week at home. Each session will last 60 minutes. The resistance training group will perform traditional resistance exercises with an intensity of 30%-60% of a voluntary repetition maximum and 1 to 2 sets of 10 repetitions each exercise. The repetitive task training group will carry out exercises involving upper and lower limbs. To determine the clinical-demographic characterization of the study population, descriptive statistics (mean and standard deviation) will be used; the correlation analysis will be performed using the Pearson or Spearman correlation coefficient; the comparison between the group of patients and the control group of healthy individuals will be performed using the t test or Mann-Whitney test; the comparison before and after the training programs will be performed using the t-test or Mann-Whitney; the comparison between groups will be performed using ANOVA; the normality test to be used will be the Shapiro-Wilk and the results will be considered significant for P<0.05. EXPECTED RESULTS: It is expected that FI-3 will present a good correlation with muscle function assessed by computerized isokinetic dynamometry and electromyography, given its reduced cost and less time spent on evaluation. It is also expected to demonstrate that repetitive task training is as efficient and safe as resistance exercises.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of polymyositis or dermatomyositis (Bohan and Peter criteria)
* age ≥18 years
* duration of disease since diagnosis for more than six months
* stable medication ≥3 months
* chronic inactive or mildly active but stable myositis for at least 3 months prior to observation
* Health Assessment Questionnaire (HAQ) ≥0.5

Exclusion Criteria:

* serious cardiac or pulmonary conditions
* severe osteoporosis
* unable to exercise
* neoplasm
* cognitive disorders
* acute or chronic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
muscle performance endurance | 2 years
  "Myositis Functional Index-3 (FI-3)"; number of repetition of each muscle group task from 0-60
computerized muscle endurance test | 2 years
  "isokinetic dynamometry"; number of repetitions of shoulder and hip flexion until exhaustion

SECONDARY OUTCOMES:
manual muscle strength test | 2 years
  "Manual Muscle Test 8"; Score from 0-10, higher scores mean a better outcome
computerized muscle strength test | 2 years
  "isokinetic dynamometry"; mean of 3 concentric peak torque of shoulder and hip flexion
cardiopulmonary capacity | 2 years
  "6-minute walk test"; greater time mean a better outcome
functional capacity | 2 years
  "Health Assessment Questionnaire"; Score from 0-3, score from 0-100, higher scores mean a worse outcome
quality of life level | 2 years
  "Medical Outcomes Short-Form Health Survey (SF-36)";Score from 0-100, higher scores mean a better outcome
disease activity by physician | 2 years
  "Physician Global Assessment (PGA)"; Score from 0-10, higher scores mean a worse outcome
disease activity by patient | 2 years
  "Subjective Global Assessment (SGA)"; Score from 0-10, higher scores mean a worse outcome
disease activity questionnaire | 2 years
  "Myositis Disease Activity Assessment Tool (MDAAT)"; This is a combined tool that captures the physician's assessment of disease activity of various organ systems using the 0-4 scale and a visual analog scale (VAS) from 0-10cm
laboratory parameters of disease activity I | 2 years
  "creatine phosphokinase"; units/L
laboratory parameters of disease activity II | 2 years
  aldolase; units/L
disease damage | 2 years
  "Myositis Damage Index (MDI)"; 10 cm visual analogue scale scores for each of the eleven individual organ systems
muscle activation | 2 years
  electromyography during shoulder and hip flexion; motor unit action potentials (MUAPs)
muscle damage | 2 years
  magnetic resonance imaging of thigh muscles; muscle damage and fatty infiltration

CONTACTS AND LOCATIONS:
Locations (1):
- Samira Tatiyama Miyamoto, PhD, Vitória, Espírito Santo, Brazil

IPD SHARING:
Plan to Share IPD: No